CLINICAL TRIAL: NCT03574129
Title: Adolescent Transition to Adult Care for HIV-infected Adolescents in Kenya
Acronym: ATTACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor, Epidemiology, Global Health, Medicine, Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001756; 1R01HD089850-01 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-06-29 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Adolescent Behavior; HIV; Transition; Adolescent Development; Disclosure
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: An adolescent transition package composed of a disclosure booklet and transition tool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescent transition package (Experimental): Adolescent transition package
  Interventions: Behavioral: Adolescent Transition Package
- Standard of care (No Intervention): Standard of care adolescent services

INTERVENTIONS:
Behavioral: Adolescent Transition Package — Clinic level intervention composed of an adolescent transition package with tools to support health care workers to disclose HIV status to adolescents and to track transition to adult care.
  Arms: Adolescent transition package

SUMMARY:
This study evaluates an adolescent transition package (ATP) to support HIV infected adolescents transitioning form pediatric/adolescent care to adult care. Ten clinics will receive the intervention and 10 will receive standard of care transition services.

DETAILED DESCRIPTION:
The Adolescent Transition Package (ATP) will include two components. The validated Namibia comic book for disclosure (to be used with children over 10 years of age) and transition booklet "Taking Charge" developed by stakeholders in Kenya.

The disclosure tool includes a cartoon book, readiness and tracking tools used in clinic and health care worker training material. The intervention progresses from incomplete to complete disclosure using a narrative about soldiers fighting the battle of infection as the rationale for taking medicine. This tool has been validated for use in Namibia.

The adapted transition toolkit includes a transition booklet, tracking tools to be used by health care workers and a readiness assessment checklist to be completed by study staff. The booklet has 4 chapters addressing key areas to support adolescents gain the knowledge and skills they need in adult care. The 4 chapters are: HIV treatment literacy, self management, communication and support.

ELIGIBILITY:
Inclusion Criteria:

* Facility leadership is willing to implement the intervention

Exclusion Criteria:

* Clinics already actively using transition or disclosure tools

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1095 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace John-Stewart, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- 20 HIV clinics in Nairobi, Homabay, Nakuru and Kajiado counties, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangale DI, Onyango A, Mugo C, Mburu C, Chhun N, Wamalwa D, Njuguna I, Means AR, John-Stewart G, Weiner BJ, Beima-Sofie K. Characterizing provider-led adaptations to mobile phone delivery of the Adolescent Transition Package (ATP) in Kenya using the Framework for Reporting Adaptations and Modifications to Evidence-based Implementation Strategies (FRAME-IS): a mixed methods approach. Implement Sci Commun. 2023 Aug 14;4(1):95. doi: 10.1186/s43058-023-00446-y. PMID 37580836
- [Derived] Mburu C, Njuguna I, Neary J, Mugo C, Moraa H, Beima-Sofie K, Onyango A, Oyiengo L, Richardson BA, John-Stewart G, Wamalwa D. Mortality and Loss to Follow-Up Among Adolescents and Young Adults Attending HIV Care Programs in Kenya. AIDS Patient Care STDS. 2023 Jul;37(7):323-331. doi: 10.1089/apc.2023.0019. PMID 37432311
- [Derived] Njuguna IN, Beima-Sofie K, Mburu CW, Mugo C, Itindi J, Onyango A, Neary J, Richardson BA, Oyiengo L, Wamalwa D, John-Stewart G. Transition to independent care for youth living with HIV: a cluster randomised clinical trial. Lancet HIV. 2022 Dec;9(12):e828-e837. doi: 10.1016/S2352-3018(22)00244-2. Epub 2022 Oct 26. PMID 36309040
- [Derived] Njuguna IN, Beima-Sofie K, Mburu CW, Mugo C, Neary J, Itindi J, Onyango A, Richardson BA, Rubin Means A, Sharma M, Weiner BJ, Wagner AD, Oyiengo L, Wamalwa D, John-Stewart G. Adolescent transition to adult care for HIV-infected adolescents in Kenya (ATTACH): study protocol for a hybrid effectiveness-implementation cluster randomised trial. BMJ Open. 2020 Dec 2;10(12):e039972. doi: 10.1136/bmjopen-2020-039972. PMID 33268417

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1095 enrolled, we have excluded 25 who did not meet age criteria for the intervention (15-24) or who withdrew consent.
Groups:
- Adolescent Transition Package: Received the study intervention
- Standard of Care: Did not receive study intervention
Period: Overall Study
Arm/Group | Adolescent Transition Package | Standard of Care
Started | 578 | 488
Completed | 506 | 440
Not Completed | 72 | 48

BASELINE CHARACTERISTICS:
Groups:
- Adolescent Transition Package: Baseline characteristics of participants in intervention arm
- Standard of Care: Baseline characteristics of participants in control arm
- Total: Total of all reporting groups
Arm/Group | Adolescent Transition Package | Standard of Care | Total
Number analyzed (Participants) | 578 | 488 | 1066
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21.1 [18.3 to 22.9] | 19.7 [17.0 to 22.5] | 20.5 [17.5 to 22.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 432 | 338 | 770
  Male | 146 | 150 | 296
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 578 | 488 | 1066
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 578 | 488 | 1066
Primary caregiver [Count of Participants; unit: Participants]
  Parent | 227 | 241 | 468
  Sibling | 49 | 28 | 77
  Grand parent | 31 | 43 | 74
  Spouse | 202 | 103 | 305
  Other | 69 | 73 | 142
Entry point [Count of Participants; unit: Participants]
  PMTCT clinics | 201 | 129 | 330
  HIV clinic | 367 | 344 | 711
  Other | 9 | 15 | 24
  missing | 1 | 0 | 1
Months since disclosure of HIV status [Median (Inter-Quartile Range); unit: months] | 34 [17 to 62] | 45 [21 to 82] | 42 [19 to 69]
Baseline Transition readiness score (overall) [Mean (Standard Deviation); unit: score on a scale] — Total scale score was 18, the higher the score the better the outcome Population: Scores are aggregate of total domain scores. Some participants did not respond to all the questions in the score.
  score on a scale
    number analyzed (Participants) | 524 | 445 | 969
    (all) | 12.1 (3.4) | 11.4 (3.7) | 11.8 (3.6)
Baseline readiness score (HIV literacy) [Mean (Standard Deviation); unit: score on a scale] — The total score was 5, the higher the score the better the outcome Population: Some participants did not respond to some of the questions that comprise the score.
  score on a scale
    number analyzed (Participants) | 565 | 477 | 1042
    (all) | 2.6 (1.5) | 2.3 (1.5) | 2.5 (1.5)
Baseline readiness score (Self-management) [Mean (Standard Deviation); unit: score on a scale] — The total score was 5, the higher the score the better the outcome Population: Some participants did not respond to some of the questions that comprise the score
  score on a scale
    number analyzed (Participants) | 558 | 472 | 1030
    (all) | 3.9 (1.0) | 3.8 (1.1) | 3.9 (1.0)
Baseline readiness score (Communication) [Mean (Standard Deviation); unit: score on a scale] — The total score was 5, the higher the score the better the outcome Population: Some participants did not respond to some of the questions that comprise the score
  score on a scale
    number analyzed (Participants) | 564 | 473 | 1037
    (all) | 3.9 (1.0) | 3.8 (1.1) | 3.9 (1.1)
Baseline readiness score (Support) [Mean (Standard Deviation); unit: score on a scale] — The total score was 3, the higher the score the better the outcome Population: Some participants did not respond to some of the questions that comprise the score
  score on a scale
    number analyzed (Participants) | 563 | 478 | 1041
    (all) | 1.7 (1.0) | 1.6 (1.0) | 1.6 (1.1)
Viral suppression at baseline [Count of Participants; unit: Participants] — Population: Viral load data not available for all enrolled participants
  Participants
    number analyzed (Participants) | 456 | 401 | 857
    (all) | 382 | 326 | 708

OUTCOME MEASURES:

1. Primary Outcome: Transition Readiness Score Overall
Description: The scale name is the "Taking Charge transition readiness assessment". The scale measures readiness to transition to adult care. The scale has questions measuring attainment of knowledge and skills to navigate adult care systems. The scale is divided into 4 domains: HIV literacy (maximum score is 5, minimum 0), self-management (maximum score is 9, minimum 0), communication (maximum score is 5, minimum is 0) and support (maximum score 3, minimum is 0). The higher the score the more prepared an adolescent is to transition to adult care. For this outcome, scores across all domains will be summed to get a total readiness score (maximum score 22, minimum 0).
Time Frame: 1 year
Population: The number of participants at month 12 are less than the number enrolled due to losses to follow-up, deaths or unanswered question items
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescent Transition Package; Standard of Care: Month 12 transition readiness score (Total score)
Arm/Group | Adolescent Transition Package | Standard of Care
Number analyzed (Participants) | 476 | 416
score on a scale | 15.7 (1.8) | 13.9 (3.3)

2. Primary Outcome: Treatment Literacy Readiness Score
Description: The scale name is the "Taking Charge transition readiness assessment". The scale measures readiness to transition to adult care. The scale has questions measuring attainment of knowledge to navigate adult care systems. The higher the score the more prepared an adolescent is to transition to adult care. For this outcome we will sum scores from the HIV literacy domain (maximum score is 5, minimum 0).
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescent Transition Package; Standard of Care: Month 12 transition readiness score (HIV literacy)
Arm/Group | Adolescent Transition Package | Standard of Care
Number analyzed (Participants) | 504 | 440
score on a scale | 4.0 (1.0) | 3.0 (1.5)

3. Primary Outcome: Self Management Readiness Score
Description: The scale name is the "Taking Charge transition readiness assessment". The scale measures readiness to transition to adult care. The scale has questions measuring attainment of knowledge and skills to navigate adult care systems. The higher the score the more prepared an adolescent is to transition to adult care. For this outcome we will sum scores from the HIV literacy domain (maximum score is 9, minimum 0).
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescent Transition Package; Standard of Care: Month 12 transition readiness score (self management)
Arm/Group | Adolescent Transition Package | Standard of Care
Number analyzed (Participants) | 487 | 423
score on a scale | 4.7 (0.4) | 4.4 (0.8)

4. Primary Outcome: Communication Readiness Score
Description: The scale name is the "Taking Charge transition readiness assessment". The scale measures readiness to transition to adult care. The scale has questions measuring attainment of skills to navigate adult care systems. The higher the score the more prepared an adolescent is to transition to adult care. For this outcome we will sum scores from the HIV literacy domain (maximum score is 5, minimum 0).
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescent Transition Package; Standard of Care: Month 12 transition readiness score (communication)
Arm/Group | Adolescent Transition Package | Standard of Care
Number analyzed (Participants) | 502 | 438
score on a scale | 4.7 (0.5) | 4.4 (0.8)

5. Primary Outcome: Support Readiness Score
Description: The scale name is the "Taking Charge transition readiness assessment". The scale measures readiness to transition to adult care. The scale has questions measuring attainment of skills to navigate adult care systems. The higher the score the more prepared an adolescent is to transition to adult care. For this outcome we will sum scores from the HIV literacy domain (maximum score is 3, minimum 0).
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescent Transition Package; Standard of Care: Month 12 transition readiness score (support)
Arm/Group | Adolescent Transition Package | Standard of Care
Number analyzed (Participants) | 500 | 438
score on a scale | 2.3 (0.8) | 2.1 (1.0)

6. Secondary Outcome: Overall Retention Among 10-24 Year Old Adolescents
Description: Proportion of 10-24 year old adolescents completing visits within 6 months of last visit
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent Transition Package; Standard of Care: Month 12 retention in study
Arm/Group | Adolescent Transition Package | Standard of Care
Number analyzed (Participants) | 543 | 454
Participants | 506 | 440

7. Secondary Outcome: Number of Participants With Viral Suppression
Description: Comparisons of time to transition specific milestones between intervention and control
Time Frame: 1 year
Population: The number of participants at month 12 are less than the number enrolled due to losses to follow-up, deaths or unavailable program level data on viral suppression
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent Transition Package; Standard of Care: Proportion with viral suppression
Arm/Group | Adolescent Transition Package | Standard of Care
Number analyzed (Participants) | 275 | 277
Participants | 249 | 255

8. Other Pre Specified Outcome: Post-transition Retention
Description: completing and adult clinic visit day after transfer to adult services and at least 1 other visit within 6 months of the adult visit (total of 2 visits)
Time Frame: 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Disclosure
Description: Time to full disclosure
Time Frame: 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Adolescents With Full Disclosure by Age 10-12, 13-15 and 16-19
Description: Proportions by age group with full disclosure
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Adolescent Transition Package; Standard of Care: Proportion with adverse event
Arm/Group | Adolescent Transition Package | Standard of Care
All-Cause Mortality (participants affected / at risk) | 8/578 | 1/488
Serious Adverse Events (participants affected / at risk) | 0/578 | 0/488
Other Adverse Events (participants affected / at risk) | 0/578 | 0/488

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT03574129/Prot_SAP_000.pdf